CLINICAL TRIAL: NCT06162585
Title: Long Term Follow-up for Subjects Who Previously Participated in the NTXMCO-002 RESTORE Study
Brief Title: Non-Interventional Long Term Follow-up Study of Participants Previously Enrolled in the RESTORE Study
Acronym: REMAIN
Status: Active, not recruiting | Type: Observational
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTXLTFU-008
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa; Retinitis; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration
Keywords: Gene Therapy; AAV Vectors; Low Vision; Intravitreal Injections; Optogenetics; Multi-Characteristic Opsin; Multi-Luminance Y Mobility Test; Multi-Luminance Shape Discrimination Test; Visual Acuity
MeSH Terms: conditions — Retinitis Pigmentosa; Retinitis; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Degeneration; Vision, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation of Participants exposed 1.2E11gc/eye of MCO-010: This is a long-term follow-up observational study of participants who previously received 1.2E11gc/eye of MCO-010. No investigational product will be administered in this study.
  Interventions: Biological: Gene Therapy product-MCO-010
- Observation of Participants exposed to 0.9E11gc/eye of MCO-010: This is a long-term follow-up observational study of participants who previously received 0.9E11gc/eye of MCO-010 No investigational product will be administered in this study.
  Interventions: Biological: Gene Therapy product-MCO-010

INTERVENTIONS:
Biological: Gene Therapy product-MCO-010 — Safety evaluation to monitor long term effects of previously injected MCO-010 in RP patients

SUMMARY:
This study will be conducted following Good Clinical Practice (GCP) and International Conference on Harmonization (ICH) guidelines. Eligible subjects will be consented to return for scheduled study visits for this study following their completion in study NTXMCO-002 (RESTORE). They will not receive a second treatment with MCO-010 (or a repeated sham injection) in this study

DETAILED DESCRIPTION:
This study is designed to follow subjects with Retinitis Pigmentosa (RP) previously enrolled in study NTXMCO-002 (RESTORE, NCT04945772). In that study, 18 of 27 enrolled subjects received MCO-010, an ambient light-activated, Multi-Characteristic Opsin (MCO) transgene in an adeno-associated virus serotype 2 (AAV2) vector via intravitreal injection (IVT) and 9 of 27 received a sham injection. Those who received the sham injection will not be continued in the long-term, follow-up study for drug safety. MCO-010 has the potential to restore vision irrespective of the underlying gene mutation, and because it is directed at bipolar retinal cells, intact photoreceptors are not required. Further details on MCO-010 and the underlying disease under investigation are included in the protocol for RESTORE and are not repeated herein.

The current study is a non-interventional long-term safety follow-up of the subjects who completed RESTORE, in accordance with FDA guidance on recipients of human gene therapy products.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in study NTXMCO-002 (RESTORE)
* Able to comprehend and give informed consent.
* Able to comply with testing and all protocol tests.
* Agree to participate for the full 3-year duration of follow-up to the best of their ability and barring any unforeseen circumstances.

Exclusion Criteria:

* Not applicable. Subjects will be included in this study and will be consented after completion of all assessments at their final RESTORE study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population will be comprised of the 18 adult subjects with advanced retinitis pigmentosa, previously dosed with MCO-010 in the RESTORE study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the long-term safety of previous treatment with a single intravitreal injection of MCO-010 | 156 weeks
  Delayed adverse events. Incidence, nature, and severity of selected adverse events (AEs); all serious adverse events (SAEs); all ocular AEs including intraocular inflammation graded through ocular exam; non-ocular AEs with a common terminology criteria for adverse events (CTCAE) grade of 3 or greater; AEs of special interest (AESIs) including new malignancies, new incidence or exacerbation of any pre-existing neurologic disorder or rheumatologic or other autoimmune disorder, new incidence of hematologic disorder or new infection regardless of suspected relatedness to treatment with MCO-010.

SECONDARY OUTCOMES:
Evaluation of long-term effects on visual acuity of previous treatment with a single intravitreal injection of MCO-010 | 156 Weeks
  Change from baseline in BCVA over time in both eyes
Evaluation of long-term effects on shape discrimination at multiple light levels of previous treatment with a single intravitreal injection with MCO-010 | 156 Weeks
  Change from baseline in multi-luminance shape discrimination test (MLSDT) scores
Evaluation of long-term effects on navigation/mobility at multiple light levels of previous treatment with a single intravitreal injection with MCO-010 | 156 Weeks
  Change from baseline in multi-luminance Y-Mobility Test (MLYMT) score
Exploration of the long-term impact of previous treatment with MCO-010 on retinal thickness and retinal anatomy | 156 Weeks
  Assessment of fundus photography and Optical Coherence Tomography (OCT) outcomes over time

OTHER OUTCOMES:
Assessment of the long-term pharmacokinetic (PK) and pharmacodynamic (PD) impact of previous treatment with MCO-010 on gene reporter expression | 156 Weeks
  PK parameters including change from baseline of fundus fluorescence intensity of reporter over time and PD correlation of gene expression with the efficacy measures in the study eye and fellow eye (selected sites)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Barone, MD, Study Director — Nanoscope Therapeutics Inc.
Locations (6):
- United States (5):
  - Nanoscope Clinical Site, Beverly Hills, California
  - Nanoscope Clinical Site, Pensacola, Florida
  - Nanoscope Clinical Site, Fargo, North Dakota
  - Nanoscope Clinical Site, Houston, Texas
  - Nanoscope Clinical Site, McAllen, Texas
- Nanoscope Clinical Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed and results are analyzed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: Within a year from the long term monitoring data availability
Access Criteria: IPD sharing access will be subject to data transfer agreement. IPD generated as part of this clinical study may be subject to patient confidentiality.